CLINICAL TRIAL: NCT00984763
Title: A Phase I/IIa Study of the Safety, Immunogenicity and Parasite Growth Inhibitory Activity of AMA1-C1/Alhydrogel® + CPG 7909, an Asexual Blood Stage Vaccine for Plasmodium Falciparum Malaria
Brief Title: A Study to Assess Safety, Immunogenicity and Parasite Growth Inhibition of an Asexual Blood Stage Vaccine for P. Falciparum Malaria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC035; NCT00605462 (obsolete NCT alias)
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Malaria
Keywords: Malaria; Vaccine
MeSH Terms: conditions — Malaria | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): AMA1-C1/Alhydrogel® + CPG 7909 vaccine given twice two months apart followed by malaria parasite challenge
  Interventions: Biological: AMA1-C1/Alhydrogel® + CPG 7909
- Group 2 (No Intervention): Control: malaria parasite challenge without prior vaccinations

INTERVENTIONS:
Biological: AMA1-C1/Alhydrogel® + CPG 7909 — A 0.55 mL dose of AMA1-C1/Alhydrogel® + CPG 7909 (corresponds to 80 µg of AMA1-C1 and 564 µg of CPG 7909)
  Arms: Group 1

SUMMARY:
Malaria is a parasite, infection with which kills over 2 million people each year. It is a major problem for those who live in endemic areas and for travellers. There is a great need for a safe effective malaria vaccine. The purpose of this study is to examine a new vaccine designed to provide immunity during the blood stage of the malaria parasite's lifecycle.

The vaccine consists of AMA1-C1 which is a mixture of two recombinant synthetic AMA1 proteins from two Plasmodium falciparum strains, Alhydrogel® which is an aluminium-based adjuvant and CPG 7909 - an oligodeoxynucleotide, which enhances immune response.

This study will enable the investigators to assess:

1. The ability of of a growth inhibition assay to predict the effectiveness of a malaria vaccine.
2. The safety of the vaccine in healthy volunteers
3. The response of the human immune system to the vaccine

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent for participation in the study
* Healthy, non pregnant adult aged 18 - 50 years
* Resident in or near Oxford for the duration of the challenge study
* Seropositive for CMV and EBV
* Female subjects of child bearing potential must be willing to ensure that they practice effective contraception during the study
* Males must be willing to use barrier contraception from day of first vaccination onwards until 3 months after the second vaccination
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study
* Agreement to permanently refrain from blood donation.

Exclusion Criteria:

* Any deviation from the normal range in biochemistry or haematology blood tests or in urine analysis as defined in Appendix B
* Female patient/subject who is pregnant, lactating or planning pregnancy during the course of the study
* Healthy volunteers who have participated in another research study involving an investigational product in the past 12 weeks
* Subjects who have previously received an investigational malaria vaccine
* History of malaria chemoprophylaxis with chloroquine within 5 months prior to the planned challenge, with Lariam within 6 weeks prior to the challenge, and Riamet® within 2 weeks prior to the challenge
* Travel to a malaria endemic area within the previous 6 months
* Planned travel to malarious areas during the study period
* Any history of malaria
* Contraindication to both anti-malarial drugs (Riamet® and chloroquine)
* concomitant use of other drugs known to cause QT-interval prolongation, ( e.g. macrolides, quinolones, amiodarone etc)
* An estimated ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system (Conroy 2003)
* Family history of sudden cardiac death
* History of cardiac arrhythmia or prolonged QT syndrome
* Any history of severe allergic reaction or anaphylaxis
* History of a known allergy to nickel
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months
* History or evidence of pre-existing autoimmune or antibody mediated disease or laboratory evidence of possible autoimmune disease (defined as anti-dsDNA ≥ 25 IU/mL)
* Seropositive for hepatitis B surface antigen (HBsAg) or antibodies to hepatitis C virus
* Any on-going chronic illness requiring hospital specialist supervision
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* History of or current intravenous drug abuse
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or may influence the result of the study, or the subject's ability to participate in the study.
* Investigator assessment of lack of willingness to participate and comply with all requirements of the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate a correlation between in vitro growth inhibition assay and parasite multiplication rate in vivo | Up to 16 days following blood stage parasite challenge

SECONDARY OUTCOMES:
To detect differences in the multiplication rate responses between unvaccinated control subjects and volunteers vaccinated with AMA1-C1/Alhydrogel® + CPG 7909 | Up to 16 days following blood stage parasite challenge

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, D.Phil, FRCP, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, Headington, United Kingdom

REFERENCES:
- [Derived] Duncan CJ, Sheehy SH, Ewer KJ, Douglas AD, Collins KA, Halstead FD, Elias SC, Lillie PJ, Rausch K, Aebig J, Miura K, Edwards NJ, Poulton ID, Hunt-Cooke A, Porter DW, Thompson FM, Rowland R, Draper SJ, Gilbert SC, Fay MP, Long CA, Zhu D, Wu Y, Martin LB, Anderson CF, Lawrie AM, Hill AV, Ellis RD. Impact on malaria parasite multiplication rates in infected volunteers of the protein-in-adjuvant vaccine AMA1-C1/Alhydrogel+CPG 7909. PLoS One. 2011;6(7):e22271. doi: 10.1371/journal.pone.0022271. Epub 2011 Jul 22. PMID 21799809